CLINICAL TRIAL: NCT03418545
Title: A Multicenter, Single-blind, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLBELLA® XC Injectable Gel for Correction of Infraorbital Hollowing
Brief Title: A Safety and Effectiveness of VOLBELLA XC Hyaluronic Acid (HA) Injectable Gel to Correct Infraorbital Hollowing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1932-701-008
Record Dates: First submitted 2018-01-17; First posted 2018-02-01 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Infraorbital Hollowing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- JUVÉDERM VOLBELLA® XC (Experimental): JUVÉDERM® VOLBELLA™ XC injectable gel was injected into the infraorbital and adjacent area at Randomization as determined by the investigator. Participants were eligible to receive an optional touch-up treatment 1 month later and an optional repeat treatment 12 months after last treatment, if applicable. A maximum of 2.2 milliliter (mL) per side was injected for initial and touch-up treatments combined.
  Interventions: Device: JUVÉDERM VOLBELLA® XC injectable gel
- No-treatment Control (No Intervention): Participants randomized to the No-treatment Control group completed a 3-month No-treatment Period. Participants were then eligible to receive optional treatment with JUVÉDERM® VOLBELLA™ XC injectable gel injected into the infraorbital and adjacent area followed by an optional touch-up treatment 1 month later.

INTERVENTIONS:
Device: JUVÉDERM VOLBELLA® XC injectable gel — JUVÉDERM® VOLBELLA™ XC dermal filler injected into the infraorbital and adjacent area.
  Arms: JUVÉDERM VOLBELLA® XC

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of JUVÉDERM® VOLBELLA™ XC in adult participants seeking correction of hollowing of the tear troughs.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 22 or over and in good general health
* Has "Moderate" or "Severe" infraorbital hollowing (grade 2 or 3 on the Allergan Infraorbital Hollows Scale (AIHS)) for each eye as assessed by the Evaluating Investigator (i.e., both eyes must qualify but do not need to have the same score)
* Is able to complete effectiveness self-assessments without the use of glasses (contact lens use is acceptable if they will be used for all subject self-assessments)
* Ability to follow study instructions and likely to complete all required visits
* Written informed consent has been obtained

EXCLUSION CRITERIA:

* Has hyperpigmentation in the infraorbital area (does not include dark circles under the eyes not due to hyperpigmentation)
* Has ever received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
* Has ever undergone fat injections above the subnasale or is planning to undergo this procedure during the study
* Has tattoos, piercings, facial hair (i.e., beard, mustache), or scars that would interfere with visual assessment of the infraorbital hollows
* Has undergone volume augmentation with semipermanent dermal fillers (e.g., calcium hydroxyapatite, poly-L-lactic acid) or temporary dermal fillers in the malar area, temples, or around the eyes within 12 months before enrollment or is planning to undergo such treatment during the study
* Has begun using any new over-the-counter or prescription oral or topical, anti-wrinkle products within 30 days before enrollment or is planning to begin using such products during the study. Subjects who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study)
* Has active or recurrent inflammation or infection in either eye
* Has active autoimmune disease
* Females who are pregnant, nursing, or planning a pregnancy
* Is an employee (or a relative of an employee) of the treating investigator (TI), evaluating investigator (EI), or Allergan, or a representative of Allergan
* Has a condition or is in a situation which in the TI's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Abrams, Study Director — Allergan
Locations (15):
- United States (15):
  - Christopher I. Zoumalan MD Inc., Beverly Hills, California
  - Steve Yoelin MD Medical Associate, Inc., Newport Beach, California
  - Cosmetic Laser Dermatology, San Diego, California
  - Facesplus, Inc., San Diego, California
  - Art of Skin MD, Solana Beach, California
  - Steven Fagien M.D.F.A.C.S., Boca Raton, Florida
  - Center For Sight, Sarasota, Florida
  - Lupo Center for Aesthetic and General Dermatology, New Orleans, Louisiana
  - Image Dermatology, P.C., Montclair, New Jersey
  - Williams Plastic Surgery Specialists, Latham, New York
  - Aesthetic Solutions, PA., Chapel Hill, North Carolina
  - Duke Aesthetic Center, Durham, North Carolina
  - Brian Biesman, MD, Nashville, Tennessee
  - Precision Dermatology, Bellaire, Texas
  - The Center for Skin Research, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. — http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 163 participants were enrolled in the study (signed the informed consent) out of which 140 were randomized to receive JUVÉDERM® VOLBELLA™ XC (treatment group) or no treatment (control group) in 3:1 ratio.
Groups:
- No-treatment Control: Participants randomized to the No-treatment Control group completed a 3-month No-treatment Period (Control Period). Participants were then eligible to receive optional treatment with JUVÉDERM® VOLBELLA™ XC injectable gel injected into the infraorbital and adjacent area followed by an optional touch-up treatment 1 month later.
- JUVÉDERM® VOLBELLA™ XC: JUVÉDERM® VOLBELLA™ XC injectable gel was injected into the infraorbital and adjacent area at Randomization as determined by the investigator. Participants were eligible to receive an optional touch-up treatment 1 month later and an optional repeat treatment 12 months after last treatment, if applicable. A maximum of 2.2 mL per side was injected for initial and touch-up treatments combined.
Period: Overall Study
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA™ XC
Started | 35 | 105
Safety Population (Safety Population included participants who were randomized to study treatment (JUVÉDERM® VOLBELLA™ XC treatment group) and received at least 1 study device treatment and participants who were randomized to the control group.) | 34 | 105
Received Optional or Repeat Treatment (Participants randomized to the No-treatment Control group who received optional treatment with JUVÉDERM® VOLBELLA™ XC injectable gel after Month 3 and participants randomized to the JUVÉDERM® VOLBELLA™ XC arm who received repeat treatment with JUVÉDERM® VOLBELLA™ XC injectable gel 12 months after the initial treatment.) | 29 | 37
Completed | 30 | 94
Not Completed | 5 | 11
Not completed — Withdrawal by Participant | 2 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Reason Not Specified | 0 | 1
Not completed — Missing Completion Status | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) Population included participants who were randomized to study treatment (JUVÉDERM® VOLBELLA™ XC treatment group), received at least 1 study device treatment and had a Baseline and at least 1 posttreatment assessment of the primary effectiveness variable and participants who were randomized to the control group and had a Baseline and at least 1 follow-up assessment of the primary effectiveness variable.
Groups:
- Total: Total of all reporting groups
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA™ XC | Total
Number analyzed (Participants) | 32 | 103 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.85) | 44.9 (10.58) | 43.9 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 93 | 124
  Male | 1 | 10 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 18
  Not Hispanic or Latino | 25 | 92 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 16 | 18
  White | 27 | 81 | 108
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 1-point Improvement Change From Baseline on the Allergan Infraorbital Hollows Scale (AIHS) Based on Evaluating Investigator's (EI) Assessment
Description: The evaluating investigator assessed hollowing in both infraorbital areas using the 5-point photonumeric AIHS where: 0=none (no visible hollowing or volume loss medially or laterally), 1=minimal (presence of hollowing with some volume loss medial to the mid-pupillary line; smooth lateral lid-cheek transition), 2=moderate (defined hollowing extending laterally beyond the mid-pupillary line with moderate volume loss; smooth lateral lid-cheek transition with mild volume loss), 3=severe (defined hollowing extending laterally beyond the mid-pupillary line with moderate volume loss creating a defined groove along the lid-cheek junction), 4=extreme (defined hollowing extends from medial to lateral canthus; severe volume loss creates a marked step along the lid-cheek junction). The percentage of participants with at least a 1-point improvement change (decrease) in the AIHS is reported.
Time Frame: Baseline (Screening) to Month 3 post last treatment (JUVÉDERM® VOLBELLA™ XC arm) or Month 3 post randomization (No-treatment Control arm)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA™ XC
Number analyzed (Participants) | 32 | 103
percentage of participants | 15.6 [3.0 to 28.2] | 83.1 [75.8 to 90.4]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLBELLA™ XC; Test type: Superiority; p < 0.0001, Fisher Exact — The p-value and 95% CI are computed by pooling 5 imputed datasets using PROC MIANALYZE in SAS with normal approximation. The p-value and 95% CI for each imputed data set is based on the Fisher's exact test and the Wald test, respectively; Percentage difference = 67.5, 95% CI 2-sided [52.9 to 82.0]

2. Secondary Outcome: Percentage of Participants Improved or Much Improved in the Overall Aesthetic Assessment Based on EI's Assessment of the Global Aesthetic Improvement Scale (GAIS) at Month 3 After the Last Treatment
Description: The evaluating investigator assessed a participant's global aesthetic improvement in the infraorbital area compared to Baseline using the 5-point GAIS where: 2=much improved (marked improvement in appearance), 1=improved (improvement in appearance, but a touch-up or retreatment is indicated), 0=no change (appearance is essentially the same as the original condition), -1=worse (appearance is worse than the original condition), -2=much worse (appearance is much worse than the original condition). The percentage of participants where the EI selected improved or much improved is reported.
Time Frame: Baseline (Randomization) to Month 3 post last treatment (JUVÉDERM® VOLBELLA™ XC) or Month 3 post randomization (No-treatment Control arm)
Population: mITT Population included participants who were randomized to study treatment (JUVÉDERM® VOLBELLA™ XC treatment group), received at least 1 study device treatment and had a Baseline and at least 1 posttreatment assessment of the primary effectiveness variable and participants who were randomized to the control group and had a Baseline and at least 1 follow-up assessment of the primary effectiveness variable. Overall number analyzed are the participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA™ XC
Number analyzed (Participants) | 32 | 100
percentage of participants | 12.5 [3.5 to 29.0] | 86.0 [77.6 to 92.1]
Statistical Analysis 1: Comparison: No-treatment Control vs JUVÉDERM® VOLBELLA™ XC; Test type: Superiority; Percentage difference = 73.5, 95% CI 2-sided [60.2 to 86.8] — The 95% CI is based on the Wald test

3. Secondary Outcome: Percentage of Participants Improved or Much Improved in the Overall Aesthetic Assessment Based on Participant's Assessment of the GAIS at Month 3 After the Last Treatment
Description: The participant assessed their global aesthetic improvement in the infraorbital area compared to Baseline using the 5-point GAIS where: 2=much improved (marked improvement in appearance), 1=improved (improvement in appearance, but a touch-up or retreatment is indicated), 0=no change (appearance is essentially the same as the original condition), -1=worse (appearance is worse than the original condition), -2=much worse (appearance is much worse than the original condition). The percentage of participants who selected improved or much improved is reported.
Time Frame: Baseline (Randomization) to Month 3 post last treatment
Population: VOLBELLA™ Initially Treated (VIT) Population included participants who were randomized and received VOLBELLA™ treatment at the beginning of the Control Period. Overall number analyzed are the participants with data available for analyses. The GAIS assessed by the participant was only completed by participants in the JUVÉDERM® VOLBELLA™ XC arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JUVÉDERM® VOLBELLA™ XC
Number analyzed (Participants) | 100
percentage of participants | 84.0 [75.3 to 90.6]

4. Secondary Outcome: Mean Change From Baseline in Rasch-Transformed Score Based on Participant Responses on the FACE-Q™ Appraisal of Lower Eyelids Questionnaire to Month 3 After the Last Treatment
Description: Participants assessed their overall satisfaction by using 7 questions on the validated Appraisal of Lower Eyelids module of the FACE-Q™ questionnaire. Each question was answered on a 4-point scale where: 1=not at all, 2=a little, 3=moderately, and 4=extremely bothered. The responses to the items were transformed to create a Rasch transformed score that ranges from 0=worst to 100=best. Higher scores indicate higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Randomization) to Month 3 post last treatment
Population: VIT Population included participants who were randomized and received VOLBELLA™ treatment at the beginning of the Control Period. Overall number analyzed are the participants with data available for analyses at Baseline. Number analyzed is the number of participants with data available for analyses at a given time point. The FACE-Q™ was only completed by participants in the JUVÉDERM® VOLBELLA™ XC arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JUVÉDERM® VOLBELLA™ XC
Number analyzed (Participants) | 104
score on a scale
  Baseline | 54.5 (14.23)
  Change From Baseline at Month 3: number analyzed (Participants) | 101
  Change From Baseline at Month 3 | 17.8 (19.80)
Statistical Analysis 1: Comparison: JUVÉDERM® VOLBELLA™ XC; Test type: Superiority; p < 0.0001, t-test, 2 sided — A 2-sided paired t-test at the 5% level was performed to demonstrate that the mean overall satisfaction score at Month 3 was statistically greater than that at Baseline for the treatment group

ADVERSE EVENTS:
Time Frame: From Randomization to the end of the study (JUVÉDERM® VOLBELLA™ XC: Up to 14 months; No-treatment Control: Up to 13 months)
Description: All-Cause Mortality: All randomized participants. Serious Adverse Events and Other Adverse Events: Safety Population included participants who were randomized to study treatment (JUVÉDERM® VOLBELLA™ XC treatment group) and received at least 1 study device treatment and participants who were randomized to the control group. The data for adverse events is added as per treatment received by the participants.
Groups:
- JUVÉDERM® VOLBELLA™ Initial Treatment: JUVÉDERM® VOLBELLA™ XC injectable gel was injected into the infraorbital and adjacent area at Randomization as determined by the investigator.
- JUVÉDERM® VOLBELLA™ Optional Treatment: Participants randomized to the No-treatment Control group received optional treatment with JUVÉDERM® VOLBELLA™ XC injectable gel, injected into the infraorbital and adjacent area Month 3 after Randomization as determined by the investigator.
- JUVÉDERM® VOLBELLA™ Repeat Treatment: Participants randomized to the JUVÉDERM® VOLBELLA™ XC arm received JUVÉDERM® VOLBELLA™ XC injectable gel injected into the infraorbital and adjacent area 12 months after the last treatment as determined by the investigator.
Arm/Group | No-treatment Control | JUVÉDERM® VOLBELLA™ Initial Treatment | JUVÉDERM® VOLBELLA™ Optional Treatment | JUVÉDERM® VOLBELLA™ Repeat Treatment
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/105 | 0/29 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/105 | 0/29 | 1/37
Other Adverse Events (participants affected / at risk) | 0/34 | 0/105 | 3/29 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (N=34) | JUVÉDERM® VOLBELLA™ Initial Treatment (N=105) | JUVÉDERM® VOLBELLA™ Optional Treatment (N=29) | JUVÉDERM® VOLBELLA™ Repeat Treatment (N=37)
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No-treatment Control (N=34) | JUVÉDERM® VOLBELLA™ Initial Treatment (N=105) | JUVÉDERM® VOLBELLA™ Optional Treatment (N=29) | JUVÉDERM® VOLBELLA™ Repeat Treatment (N=37)
Injection site bruising (General disorders) | 0 | 0 | 2 | 0
Injection site swelling (General disorders) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT03418545/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03418545/SAP_001.pdf